CLINICAL TRIAL: NCT07094763
Title: Efficacy and Safety of Tenecteplase Intravenous Thrombolysis in Acute Posterior Circulation Ischemic Stroke Within 4.5-24 Hours After Onset: A Multicenter, Prospective, Randomized, Open-Label, Blinded Endpoint Trial
Brief Title: Efficacy and Safety of Tenecteplase Intravenous Thrombolysis in Acute Posterior Circulation Ischemic Stroke Within 4.5-24 Hours After Onset
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Attention-Extend IV
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
Keywords: TNK Intravenous Thrombolysis; Acute ischemic stroke; posterior circulation; Beyond optimal time window
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard medical management (Active Comparator): standard medical management
  Interventions: Drug: standard medical management
- TNK plus standard medical treatment (Experimental): Patients in the TNK treatment group will receive TNK intravenous thrombolysis and the usual dosage for TNK intravenous thrombolysis is 0.25mg/Kg, with a maximum of 25mg.
  Interventions: Drug: TNK plus standard medical treatment

INTERVENTIONS:
Drug: TNK plus standard medical treatment — Patients in the TNK treatment group will receive TNK intravenous thrombolysis and the usual dosage for TNK intravenous thrombolysis is 0.25mg/Kg, with a maximum of 25mg.
  Arms: TNK plus standard medical treatment
Drug: standard medical management — standard medical management
  Arms: standard medical management

SUMMARY:
This study aims to evaluate the efficacy and safety of tenecteplase (TNK) intravenous thrombolysis within the extended time window (4.5 to 24 hours) in patients with acute posterior circulation ischemic stroke.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, controlled trial assesses the efficacy and safety of intravenous tenecteplase for acute posterior-circulation ischemic stroke treated 4.5-24 hours after onset. Participants with imaging-confirmed stroke will be randomly assigned 1:1 to receive either tenecteplase or standard medical therapy. Eligible patients must present within 4.5-24 hours from symptom onset, defined as the midpoint between last known normal and first observed neurological deficit. All participants will undergo telephone follow-up at 3 months and 1 year, with the modified Rankin Scale as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Meeting at least one of the following criteria: acute posterior circulation ischemic stroke confirmed by MRI; symptomatic stenosis or occlusion of a posterior circulation large vessel on vascular imaging (CTA/MRA/DSA); perfusion imaging demonstrating clinically relevant hypoperfusion in the posterior circulation territory.
3. Onset time between 4.5-24 hours (for wake-up stroke or unwitnessed stroke, onset time is defined as the midpoint between last known well and symptom detection).
4. NIHSS score>3.
5. PC-ASPECTS ≥7 (if discrepancy exists between DWI and CT findings, CT assessment takes precedence).
6. Pre-stroke mRS ≤1.
7. Signed informed consent by the patient or legally authorized representative.

Exclusion Criteria:

1. Contraindication to tenecteplase or its components.
2. Planing to receive endovascular therapy with thrombectomy, angioplasty or stenting whin 3 months.
3. Acute anterior circulation infarction confirmed by MRI, anterior circulation large vessel occlusion on vascular imaging (CTA/MRA/DSA), or anterior circulation hypoperfusion on perfusion imaging.
4. History of intracranial hemorrhage.
5. Stroke, myocardial infarction, severe traumatic brain injury, or intracranial/spinal surgery within the preceding 3 months.
6. Intracranial tumor, arteriovenous malformation (AVM), or giant aneurysm.
7. Active internal bleeding, major surgery, trauma, gastrointestinal/urinary tract bleeding within 3 weeks.
8. Non-compressible arterial puncture within 1 week.
9. Suspected aortic dissection.
10. Clinically significant bleeding or coagulopathy, including: Warfarin use with INR >1.7 or PT >15 s; Low-molecular-weight heparin within 24 hours; Direct oral anticoagulants within 48 hours; Laboratory abnormalities (e.g., APTT >40 s).
11. Platelet dysfunction or platelet count <100×10⁹/L.
12. Uncontrolled hypertension (systolic BP >180 mmHg or diastolic BP >110 mmHg unresponsive to antihypertensive therapy).
13. Uncontrolled hypoglycemia/hyperglycemia (<50 mg/dL [2.8 mmol/L] or >400 mg/dL [22.2 mmol/L]).
14. Pregnancy or lactation.
15. A life expectancy of less than three months.
16. Participation in other clinical trials within 3 months or ongoing trial enrollment.
17. Inability to follow up (e.g., no fixed residence, overseas patients).
18. Patient deemed unsuitable for the trial by site investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Scale (mRS) score 0-1 at 90 ±14 days; | 90 ±14 days

SECONDARY OUTCOMES:
Proportion of patients with mRS score 0-2 at 90 ±14 days; | 90 ±14 days
Proportion of patients with mRS score 0-3 at 90 ±14 days; | 90 ±14 days
Ordinal distribution of mRS score at 90 ±14 days; | 90 ±14 days
Change in NIHSS score at 24-36 hours post-treatment | 24 hours post-treatment
5)Change in NIHSS score at 5-7 days post-treatment; | 5-7 days post-treatment
EQ-5D-5L questionnaire score at 90 ±14 days; | 90 ±14 days
Barthel Index score at 90 ±14 days; | 90 ±14 days
1)Symptomatic intracranial hemorrhage within 36 hours (Heidelberg criteria) | 24-36 hours after treatment
Any intracranial hemorrhage within 36 hours (Heidelberg criteria) | 24-36 hours after treatment
Mortality rate at 90 ±14 days | 90 ±14 days
Overall incidence of serious adverse events | 90 ±14 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of the University of Science and Technology of China, Hefei, China

IPD SHARING:
Plan to Share IPD: No